CLINICAL TRIAL: NCT06085703
Title: A Prospective, Randomized, Open Label, Parallel, 6-month Study to Explore and Evaluate the Therapeutic Effects of Henagliflozin on the Cognitive Function, Olfactory Function, and Odor-induced Brain Activation in T2DM Patients With Mild Cognitive Impairment.
Brief Title: Effects of Henagliflozin on the Brain Function in T2DM Patients With Mild Cognitive Impairment: a Randomized, Parallel Controlled Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Zhu DaLong, Chief Physician, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ZZ2023
Record Dates: First submitted 2023-10-10; First posted 2023-10-17 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2023-10

CONDITIONS: Type 2 Diabetes Mellitus; Mild Cognitive Impairment
Keywords: Functional MRI; Cognition; Olfactory function; Henagliflozin and Gliclazide
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Cognitive Dysfunction | interventions — henagliflozin; Metformin; Gliclazide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Henagliflozin Group (Experimental): Henagliflozin will be initiated and maintained at 5mg/ day every morning until the completion of the study. Meanwhile, all patients will also continue on their existing dose and regimen of metformin throughout the study. Visits at 8-week intervals will be performed to evaluate the safety of drugs. Metformin dose can be reduced in response to hypoglycaemia, but Empagliflozin could not be adjusted. If the plasma glucose still not achieve the target at the maximum dose, the maximum dose will be maintained until the completion of the study.
  Interventions: Drug: Henagliflozin
- Gliclazide Group (Experimental): Gliclazide will be initiated and maintained at 30mg/ day every morning until the completion of the study. Meanwhile, all patients will also continue on their existing dose and regimen of metformin throughout the study. Visits at 8-week intervals will be performed to evaluate the safety of drugs. Metformin dose can be reduced in response to hypoglycaemia, but Gliclazide could not be adjusted. If the plasma glucose still not achieve the target at the maximum dose, the maximum dose will be maintained until the completion of the study.
  Interventions: Drug: Gliclazide

INTERVENTIONS:
Drug: Henagliflozin — Henagliflozin will be initiated and maintained at 5mg/day every morning. If necessary, the dose can be increased to 10mg once daily. All patients will also continue on their existing dose and regimen of metformin throughout the study.
  Other Names: metformin
  Arms: Henagliflozin Group
Drug: Gliclazide — Gliclazide will be initiated and maintained at 30mg/day every morning. If necessary, the dose can be increased to 120mg once daily. All patients will also continue on their existing dose and regimen of metformin throughout the study.
  Other Names: metformin
  Arms: Gliclazide Group

SUMMARY:
This is a prospective, randomized, open label, parallel, 16-week study to explore and evaluate the therapeutic effects of Henagliflozin on the cognitive function, olfactory function, and odor-induced brain activation in T2DM patients with mild cognitive impairment (MCI).

DETAILED DESCRIPTION:
This is a prospective, randomized, open label, parallel, 16-week study to explore and evaluate the therapeutic effects of Henagliflozin on the cognitive function, olfactory function, and odor-induced brain activation in T2DM patients with MCI inadequately controlled with metformin monotherapy. The control group was treated with Gliclazide. We have 1 principal investigator, 6 sub-investigators and 1 nurse in research centre. The sub-investigators will screen in the outpatient and inpatient departments to enroll 24 patients (12 patients for each arm) totally with the inclusion and exclusion criteria. The patients will be randomized at a 1:1 ratio into Henagliflozin and Gliclazide treatment group with a computer-generated random order. All patients will also continue on their existing dose and regimen of metformin throughout the study. At the baseline, clinical information collection, 100g-steamed bread meal test, biochemical measurement, body composition analysis, cognitive assessment, olfactory test and functional magnetic resonance imaging(fMRI) scan will be conducted for all patients. During the treatment period, visits at 8-week intervals will be performed to evaluate the safety of drugs and adjust the dose of metformin if hypoglycaemia occurs; meanwhile, fasting and 2-hour postprandial plasma glucose assayed by fingerstick, physical examination, and olfactory test will be conducted. At the end of the study, all of the assessments will be performed again for all recruited subjects, including early withdrawal patients.

ELIGIBILITY:
Inclusion Criteria:

* patients with type 2 diabetes mellitus ;
* Aged: 55 - 75 years ;
* Cognitive function assessment suggests mild cognitive impairment;
* A stable glucose-lowering regimen include Metformin alone or in combination with antidiabetic drugs other than SGLT2 inhibitors or sulfonylureas/glinides, or basic insulin for more than 2 months, and the dose of metformin≥1.0g/d;
* HbA1c: 7 - 10%;
* ≥6 years of education;
* Right-handed.

Exclusion Criteria:

* Cognitive function assessment suggests normal cognition or dementia;
* Other dementia related neurological diseases or depression, Mental dysplasia, mania, schizophrenia, etc in the past 2 years; Central nervous system diseases, including brain trauma, intracranial hemorrhage, acute cerebral infarction, etc;
* Severe sinusitis, nasal cavity and sinus polyps, skull base or nasopharyngeal tumors and other space occupying lesions;
* Congenital diseases and traumatic history of nose, maxillofacial and skull base affecting olfaction.
* With symptoms of upper respiratory tract infection, including nasal congestion, runny nose, fever, etc. on the day of MR examination;
* Diabetic Acute and chronic complications, including diabetic ketoacidosis, diabetic ketoacidosis; a hyperglycemic hyperosmolar state or severe hypoglycemic coma, etc.
* Severe impairment of heart, liver, kidney and other organs;
* Contraindications of MRI examination, such as implantation of metal prosthesis in vivo, claustrophobia, etc;
* Pregnant and lactating women;
* Receive other test drugs currently or within 3 months before participating in the project;
* Known or suspected allergic history to the test drug or similar drugs; SGLT2 inhibitor and sulfonylureas/glinides were used in recent 3 months.

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Change of olfactory brain activation by fMRI | from baseline to 16-week follow-up
  Whether the activation degree of olfactory task fMRI brain area in the two groups after intervention was different from that before treatment and the difference of changes between the two groups. All patients underwent odor-induced task fMRI on a 3.0T MR scanner with 222 volumes for task fMRI and 230 volumes for resting-state fMRI. The odor-induced task consisted of "fresh air" "rest" and "scent". Odor-induced brain activation was assessed by a general linear model using Statistical Parametric Mapping 12 (SPM12) software. Following extraction of the three separate conditions "fresh air," "scent," and "rest" from the whole sequence, contrasts were made for each participant between "fresh air > rest" and "scent > rest." Odor-induced fMRI data were analyzed in the mask of the olfactory network, including the regions of bilateral parahippocampus, amygdala, piriform cortex, insula, orbitofrontal cortex, hippocampus, and entorhinal cortices.

SECONDARY OUTCOMES:
Change of cognitive function | from baseline to 16-week follow-up
  Type 2 diabetes mellitus patients with MCI were relieved of mild cognitive impairment , which means MoCA scores were not less than 26 points after treatment, or improved referring to the MoCA score or the RBANS total score increased by 0.5 standard deviation compared with baseline after treatment.
Olfactory threshold test | from baseline to 16-week follow-up
  Whether the scores of olfactory threshold of the two groups after intervention were higher than those before treatment and the difference of changes between the two groups. Olfactory testing was performed using Olfactory Function Assessment by Computerized Testing (OLFACT) (Osmic Enterprises, Inc.). Based on the University of Pennsylvania Smell Identification Test (UPSIT), OLFACT tests were computerized, standardized, and self-administered. Threshold testing was performed by a series of binary dilutions of n-butanol solution in light mineral oil, and scores ranged from 1 to 13.5. Higher scores indicated better ability to detect odors.
Change of metabolism | from baseline to 16-week follow-up
  The changes of glycosylated hemoglobin among the two groups before and after intervention. The level of glycosylated hemoglobin <7% means better glucose metabolism.

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Endocrinology, the Affiliated Drum Tower Hospital of Nanjing University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zhang Z, Zhang B, Wang X, Zhang X, Yang QX, Qing Z, Zhang W, Zhu D, Bi Y. Olfactory Dysfunction Mediates Adiposity in Cognitive Impairment of Type 2 Diabetes: Insights From Clinical and Functional Neuroimaging Studies. Diabetes Care. 2019 Jul;42(7):1274-1283. doi: 10.2337/dc18-2584. Epub 2019 May 21. PMID 31221697
- [Background] Zhang Z, Zhang B, Wang X, Zhang X, Yang QX, Qing Z, Lu J, Bi Y, Zhu D. Altered Odor-Induced Brain Activity as an Early Manifestation of Cognitive Decline in Patients With Type 2 Diabetes. Diabetes. 2018 May;67(5):994-1006. doi: 10.2337/db17-1274. Epub 2018 Mar 2. PMID 29500313
- [Background] Cheng H, Zhang Z, Zhang B, Zhang W, Wang J, Ni W, Miao Y, Liu J, Bi Y. Enhancement of Impaired Olfactory Neural Activation and Cognitive Capacity by Liraglutide, but Not Dapagliflozin or Acarbose, in Patients With Type 2 Diabetes: A 16-Week Randomized Parallel Comparative Study. Diabetes Care. 2022 May 1;45(5):1201-1210. doi: 10.2337/dc21-2064. PMID 35263425